CLINICAL TRIAL: NCT03441893
Title: Role of Intestinal Protozoa and Helminths in the Course of Ulcerative Colitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan (Other Government)
Responsible Party: Principal Investigator, Svetlana Osipova, MD, PhD, DS, MD, PhD, DS, Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #15.21.2
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis Exacerbation; Protozoan Infections; Helminth Infection
Keywords: ulcerative colitis, helminths, intestinal protozoan, nitazoxanide
MeSH Terms: conditions — Colitis, Ulcerative; Protozoan Infections; Trematode Infections | interventions — nitazoxanide; Tablets; Mesalamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Patients with ulcerative colitis (Active Comparator): Patients with ulcerative colitis in this group will take nitazoxanide per os
  Interventions: Diagnostic Test: parasitological diagnostics (coproscopy); Drug: Nitazoxanide 500Mg Oral Tablet
- Participants (control group) (No Intervention): only parasitological diagnostics will be performed in this group to compare the prevalence of some representatives of the microbiota
- UC patients (cohort 1) (Active Comparator): Patients with ulcerative colitis in this group will take standart therapy (mesalazin)
  Interventions: Diagnostic Test: parasitological diagnostics (coproscopy); Drug: Mesalazine 250Mg
- UC patients (cohort 2) (Placebo Comparator): Patients with ulcerative colitis in this group will take placebo tabletes
  Interventions: Diagnostic Test: parasitological diagnostics (coproscopy); Drug: Placebo tabletes
- UC patients (cohort 3) (Active Comparator): Patients with ulcerative colitis in this group will take combination standart therapy with nitazoxanide
  Interventions: Diagnostic Test: parasitological diagnostics (coproscopy); Drug: Mesalazine 250Mg Tablet and nitazoxanide 500Mg Oral Tablet

INTERVENTIONS:
Diagnostic Test: parasitological diagnostics (coproscopy) — Three stool samples for parasitological examination will be taken from ulcerative colitis patients at 1-2 days interval.
  Arms: Patients with ulcerative colitis; UC patients (cohort 1); UC patients (cohort 2); UC patients (cohort 3)
Drug: Nitazoxanide 500Mg Oral Tablet — Tab. nitazoxanide by a 1.0 g/day (two pills) twice over orally for 14 consecutive days
  Arms: Patients with ulcerative colitis
Drug: Mesalazine 250Mg Tablet and nitazoxanide 500Mg Oral Tablet — Tab. nitazoxanide by a 1.0 g/day (one pill - 500 mg) twice over orally and mesalazine 1.5 g/day (one pill - 500 mg) three times a day orally for 14 consecutive days
  Arms: UC patients (cohort 3)
Drug: Mesalazine 250Mg — Tab. mesalazine ≥3 g/day (one pill - 500 mg) three times a day orally for 14 consecutive days
  Arms: UC patients (cohort 1)
Drug: Placebo tabletes — Tab. Placebo (shugar pills) will be given to the participants
  Arms: UC patients (cohort 2)

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory disorder of the gastrointestinal tract of unknown etiology. UC is characterized by recurring episodes of inflammation limited to mucosal and submucosal layers of the colon. The object of the present study was to determine the prevalence of intestinal protozoa and helminthes in UC patients, and the role of this changes in aetiopathogenesis of diseases. Patients will be examined before and after therapy. Parasites and protozoa prevalence and intensity will be detected by triple coproscopy.Microbiological study will be conducted before therapy for detection pathogenic bacteria only from UC patients infected with B. hominis . If intestinal pathogenic bacteria are found, participants will be excluded from further investigation.

DETAILED DESCRIPTION:
The prospective cohort and randomized, double-blind, placebo controlled study will be conducted on the basis of Research Institute of Epidemiology, Microbiology and Infectious Diseases and Coloproctology department of the Republic clinical hospital №1, Ministry of Public Health of the Republic of Uzbekistan.

Participants Diagnosis of UC will be confirmed using standard clinical, endoscopic, radiographic, and pathological criteria according to the Montreal classification of extent and severity of ulcerative colitis (Silverberg MS et al. 2006). UC categories include proctitis, left-sided colitis, and extensive colitis or pancolitis. Activity of the disease will be measured by Mayo Clinic score that consists of 4 items: stool frequency, rectal bleeding, findings of flexible proctosigmoidoscopy, and patient's functional assessment (D'Haens G et al. 2007). The disease duration will be measured in years from the first time of symptoms onset.

UC patients hospitalized in coloproctology department of Republic clinical hospital №1 will be examined before surgery and receiving of medications. Additional cohort groups: the 1st one will include UC patients infected with B. hominis which will be examined before and after taking nitazoxanide (monotherapy), the 2nd group will include UC patients infected with B. hominis before and after taking nitazoxanide and mesalazine (combination therapy) and 3rd one - patients with UC infected with B. hominis before and after taking mesalazine (monotherapy).

The control group will include residents of Tashkent region without any complaints from the gastrointestinal tract, who will apply to the clinic for planned medical examinations. Suggested age of the population from 17 to 90 years

Exclusion criteria Patients with diagnosis of Crohn's disease will be excluded from the analysis. Other exclusion criteria are toxic megacolon, abdominal abscess, symptomatic colonic stricture, stoma, a history of colectomy, an increased risk of infectious complications (e.g. as a result of recent pyogenic infection, enteric pathogens detected in microbiological stool analysis, active or latent tuberculosis, immunodeficiency, hepatitis B or C, or recent live vaccination), clinically meaningful laboratory abnormalities, pregnancy or lactation, unstable or uncontrolled medical disorders, an anticipated requirements for major surgery, colonic dysplasia or adenomas, and malignant neoplasms.

For additional groups except the above mentioned the followed patients will be excluded: individuals who were operated, ever used immunosuppressants or biological drugs, infected with intestinal pathologenic bacteria, including Clostridium difficile, Salmonella spp, Shigella spp, Campylobacter spp, Yersinia spp, and Mycobacteria.

Parasitological method Collection of stool samples. Three stool samples for parasitological examination will be taken from both control subjects and UC patients at 2 days interval before therapy (all participants) and in the 2nd week of monotherapy therapy with nitazoxanide, nitazoxanide in combination with mesalazine and monotherapy with mesalazine and in 6th and 12th weeks from beginning of the therapy. Stool samples (1-2g.) will be collected in individual containers, with 5 ml of Turdiev's preservative provided conservation and staining of proozoa cysts and eggs of worms for a year. The Turdiev's preservative includes: 80 ml of 0.2% aqueous solution of sodium nitrite, 10 ml of formaldehyde, 2 ml of glycerin, 8 ml of Lugol's solution, 250 ml of distilled water.

Stool samples (1-2g.) for detection of C. parvum (Cryptosporidium parvum) will be collected in individual empty containers no less 1 hour before parasitological examination.

Microscopy. Parasitological diagnosis will be performed by triple coproscopy using formalin - ethyl acetate concentration technique [Truant AL, Elliott SH] and iodine stained smears [King M.]. For preparations staining Lugol's solution will be used. The intensity of protozoa will be estimated by the number of protozoa in the field of view (ocular x10, objective x40) in iodine stained smears taken before application of formalin - ethyl acetate concentration technique, the number of protozoa will be calculated at least in 10 fields of view. 1-2, 3-4 and 5-6 microorganisms in a field of view were considered as infection of low, mean and high intensity respectively. For detection of C. parvum modified Ziehl - Neelsen method [Henricksen SA, Pohlenz JF] will be used for staining the preparations. The stained smears will be scanned with ×100 oil immersion lens for the presence of C. parvum.

Microbiological methods Microbiological methods wil be conducted for detection pathogenic bacteria, including Clostridium difficile, Salmonella spp, Shigella spp, Campylobacter spp, Yersinia spp, and Mycobacteria only from UC patients infected with B. hominis before therapy. If intestinal pathogenic bacteria are detected participants will be excluded from further investigation.

Collection of stool samples. Fecal samples will be collected from UC patients infected with B. hominis before therapy in sterile, wide-mouth, screw capped containers and immediately transferred to the laboratory, preferably within 2 h. Specimens will be processed for microscopy, anaerobic and aerobic culture, and ELISA (only for Clostridium difficile).

Procedures Parasitological examination in UC patients and population will be provided. Additional UC patients infected with B. hominis will be divided into 3 cohorts, in double-blinded fashion, to receive 1 of the following treatments: (1) patients with UC infected with B. hominis will be treated with nitazoxanide, 1.0 g/daily (two pills) twice over orally for 14 consecutive days; (2) UC patients infected with B. hominis will be treated with nitazoxanide by a 1.0 g/day (one pill - 500 mg) twice over orally and mesalazine 1.5 g/day (one pill - 500 mg) three times a day orally for 14 consecutive days; (3) patients with UC infected B. hominis will be treated with mesalazine ≥3 g/day (one pill - 500 mg) three times a day orally for 14 consecutive days. Except drugs patients of all three groups adhered to the diet. The purpose of follow-up was to monitor compliance with medications and to record response to therapy, adverse events, and recurrence of symptoms.

Other detected pathogenic protozoan and helminthes was treated by standard dosage of antiparasitic drugs.

Follow-up The study was conducted in two stages. At the first stage parasitological examination of patients with UC before treatment and population will be provided . At the second stage of the study in patients with UC infected with B. hominis drugs with anti Blastocystis activity will be applied as well as monitoring of therapy efficiency. Parasitological, microbiological, clinical and endoscopic examination will be conducted before therapy and at the 2nd, 6th and 12th weeks. At each visit, a Mayo Clinic score will be calculated and intensity/elimination of B. hominis will be determined.

Outcome measures The outcome measures of therapy are : eradication/ reduction of intensity of B. hominis infection and a clinical response of UC patients at the 2nd, 6th and 12th weeks will be defined as a reduction in the Mayo Clinic score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulcerative colitis before therapy and surgery
* Residents of Tashkent region which does not have any complaints from the gastrointestinal tract (control group)

Exclusion Criteria:

* Patients with a diagnosis of Crohn's disease
* Patients with a toxic megacolon,
* Patients with a abdominal abscess, -
* Patients with a symptomatic colonic stricture,
* Patients with a stoma,
* Patients with a a history of colectomy,
* An increased risk of infectious complications (e.g. as a result of recent pyogenic infection, enteric pathogens detected on stool analysis, active or latent tuberculosis, immunodeficiency, hepatitis B or C, or recent live vaccination),
* Clinically meaningful laboratory abnormalities,
* Pregnancy or lactation,
* An unstable or uncontrolled medical disorder,
* An anticipated requirement for major surgery,
* Colonic dysplasia or adenomas,
* Malignant neoplasms.
* Patients which operated,
* Ever used immunosuppressants or biological drugs
* In the presence of pathologic bacteria in gut microbiota, including Clostridium difficile, Salmonella spp, Shigella spp, Campylobacter spp, Yersinia spp, and Mycobacteria.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of intestinal helminths in patients with ulcerative colitis and association with pathogenesis. | up to 36 months
  In this study we expect to find intestinal helminths in patients with ulcerative colitis and determine their role in the development and course of ulcerative colitis
Prevalence of Lamblia intestinalis and Cryptosporidium parvum in patients with ulcerative colitis and association with pathogenesis | up to 36 months
  In this study we expect to find pathogenic protozoa in patients with ulcerative colitis and determine their role in the development of ulcerative colitis
Prevalence of intestinal protozoa (commensals) in patients with ulcerative colitis and association with pathogenesis | up to 36 months
  In this study we are going to determine their prevalence and role in the development of ulcerative colitis
Efficiency of antiparasitic therapy with nitazoxanide in ulcerative colitis patients infected with B. hominis | up to 24 months
  Reduction of intensity or eradication of B. hominis in stool samples of patients with ulcerative colitis
Efficiency of combination therapy with nitazoxanide and mesalazine in ulcerative colitis patients infected with B. hominis | up to 24 months
  Reduction of intensity or eradication of B. hominis in stool samples of patients with ulcerative colitis
Efficiency of monotherapy with mesalazine in ulcerative colitis patients infected with B. hominis | up to 24 months
  Reduction of intensity or eradication of B. hominis in stool samples of patients with ulcerative colitis
Clinical efficiency of antiparasitic therapy with nitazoxanide in ulcerative colitis patients infected with B. hominis | up to 24 months
  A positive/negative clinical response of disease in ulcerative colitis patients
Clinical efficiency of combination therapy with nitazoxanide and mesalazine in ulcerative colitis patients infected with B. hominis | up to 24 months
  A positive/negative clinical response of disease in ulcerative colitis patients
Clinical efficiency of monotherapy with mesalazine in ulcerative colitis patients infected with B. hominis | up to 24 months
  A positive/negative clinical response of disease in ulcerative colitis patients

REFERENCES:
- [Result] Toychiev A, Navruzov B, Pazylova D, Davis N, Badalova N, Osipova S. Intestinal protozoa and helminths in ulcerative colitis and the influence of anti-parasitic therapy on the course of the disease. Acta Trop. 2021 Jan;213:105755. doi: 10.1016/j.actatropica.2020.105755. Epub 2020 Nov 11. PMID 33188747
- See also: Article in Pubmed — https://pubmed.ncbi.nlm.nih.gov/33188747/